CLINICAL TRIAL: NCT06879275
Title: Incidence of Body Dysmorphic Disorder (BDD) in a Population of Patients Undergoing Orthognathic Surgery: a Prospective Study
Brief Title: Incidence of Body Dysmorphic Disorder (BDD) in a Population of Patients Undergoing Orthognathic Surgery
Acronym: IBDOS
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7033
Record Dates: First submitted 2025-01-21; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-01

CONDITIONS: Orthognathic Surgical Procedures; Psychiatric Disorders; Prognathism
Keywords: orthognatic surgery; body dismorphic disorder; prognathism; aesthetic surgery
MeSH Terms: conditions — Mental Disorders; Prognathism | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaire and Physical Exam — 2 self administered questionnaire for diagnosis of dismorphophobia will be administered

SUMMARY:
Assessment of the incidence of Body dismorphic disorder in a population candidated to orthognathic surgery

DETAILED DESCRIPTION:
Assessment of the incidence of Body dismorphic disorder in a population candidated to orthognathic surgery by using 3 validated questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients who are candidates for orthognathic surgery
* Age: 18 to 50 years;
* Informed consent

Exclusion Criteria:

* - Patients diagnosed with another psychiatric pathology
* Patients affected by syndromes involving the cervical-facial district
* Patients affected by clefts
* Patients affected by OSAS and candidates for orthognathic surgery for this indication
* Patients affected by connective tissue disorders (e.g. Ehler-Danlos, scleroderma, etc.)
* Patients candidates for orthognathic surgery due to facial trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: candidates to orthognathic surgery
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
primary outcomes | 2 years
  - Prevalence of body image disturbance (BDD) among patients undergoing orthognathic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Moro, MD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCSS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No